CLINICAL TRIAL: NCT02014389
Title: Objective Perimetry in Normal Subjects,Glaucoma Patients and Retinal Dystrophy Patients
Brief Title: Evaluation of Objective Perimetry Using Chromatic Multifocal Pupillometer
Status: Recruiting | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ygal Rotenstreich, Head of Electrophisiology Unit, Maurice and Gabriela Goldschleger Eye Research Institute, Sheba Medical Center
Other Study IDs: SHEBA -13 -0640-YR-CTIL
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Retinal Dystrophies; Retinitis Pigmentosa; Glaucoma
Keywords: Retinal Dystrophies; Retinitis Pigmentosa; Glaucoma; Visual Field
MeSH Terms: conditions — Retinal Dystrophies; Retinitis Pigmentosa; Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy subjects: Healthy subjects will be used as control group
- Patients: Patients with Glaucoma , Patients with retinal dystrophy

SUMMARY:
Objective perimetry can better monitor visual field defects in retinal dystrophy and Glaucoma patients than conventional subjective perimetry. The PLR ( Pupil Light Reflex to short and long wavelength stimuli should be significantly lower compared to healthy participants in areas of visual field defects in retinal dystrophy and Glaucoma patients.

DETAILED DESCRIPTION:
Pupil light reflex (PLR) will be measured by a chromatic multifocal pupillometer in response to short and long wavelength light with small spot stimulus in 76 points of the 30 degree visual field.

A computerized infrared video pupillometer will be used to record changes in pupil diameter in response to short- and long-wavelength stimuli (peak 485 nm and 620 nm, respectively) presented by 76 LEDs, 1.8mm spot size, at light intensities of 10-3000 cd/m2 and duration of 1-3 sec at different points of the 30 degree visual field

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old.
* Signing informed consent.
* Pupillary reflex to light.

Exclusion Criteria:

1. Cloudy corneas.
2. Surgical intraocular ophthalmic procedure within the past 30 days.
3. No reactive pupils.
4. Synechia of the iris to the lens after surgery or inflammation.
5. Neovascularization.
6. Axenfeld-Rieger Syndrome.
7. Iris atrophy (ICE syndrome).
8. Iris coloboma.
9. Sphincter damage due to ischemia.
10. Sphincter damage due to trauma (tears of sphincter or diffuse damage to muscle).
11. Sphincter damage due to Herpes Zoster Uveitis.
12. Sphincter damage due to high intraocular pressure.
13. Iris tumor or cyst.
14. Ectropion uvae.
15. Adie's pupil.
16. Third nerve aberrant regeneration of the iris sphincter.
17. RP patients with Optic neuropathy with the potential of producing a positive RAPD (Relative Afferent Pupillary Defect).
18. Chronic use of myotics or mydriatics.
19. Systemic medication that have affect on pupillary reflex .
20. Any condition preventing accurate measurement or examination of the pupil.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two Groups: 1. Control, 2. Patients - Glaucoma patients with early damage (nasal step) of Humphrey visual field (HVF), Glaucoma patients with advanced damage of HVF (arcuate , tubular vision) and retinal dystrophy patientsl
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PLR response amplitude and latency | single visit

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Skaat A, Sher I, Kolker A, Elyasiv S, Rosenfeld E, Mhajna M, Melamed S, Belkin M, Rotenstreich Y. Pupillometer-based objective chromatic perimetry in normal eyes and patients with retinal photoreceptor dystrophies. Invest Ophthalmol Vis Sci. 2013 Apr 17;54(4):2761-70. doi: 10.1167/iovs.12-11127. PMID 23482470